CLINICAL TRIAL: NCT07306507
Title: Comparison of vNOTES and Conventional Laparoscopic Hysterectomy: A Randomized Controlled Study of Pain, Opioid Use, and Quality of Recovery
Brief Title: vNOTES vs Laparoscopic Hysterectomy: Randomized Trial on Pain and Recovery"
Acronym: VNOTES-TLH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Fatma Acil,MD, Principal Investigator, Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11/7/2025-705
Record Dates: First submitted 2025-12-02; First posted 2025-12-29 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Hysterectomy
Keywords: vNOTES; Total Laparoscopic Hysterectomy; Postoperative Pain; Enhanced Recovery
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1 ratio to undergo either vNOTES hysterectomy or conventional total laparoscopic hysterectomy. Each participant receives only one of the two surgical interventions, and both groups are followed in parallel for outcome assessment.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigators responsible for postoperative data collection and analysis and outcome assessors were blinded to group allocation. These investigators were not involved in the surgical or anesthetic management of the patients. Due to the nature of the surgical procedures, blinding of participants and care providers was not feasible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vNOTES Group (Experimental): Patients undergo vaginal natural orifice transluminal endoscopic hysterectomy (vNOTES) using a transvaginal access port with a maximum pneumoperitoneum pressure not exceeding 15 mmHg.
  Interventions: Procedure: vNOTES Hysterectomy
- TLH Group (Active Comparator): Patients undergo conventional total laparoscopic hysterectomy using a camera port and accessory trocars from the umbilicus, and pneumoperitoneum is maintained at a pressure not exceeding 15 mmHg.
  Interventions: Procedure: Total Laparoscopic Hysterectomy

INTERVENTIONS:
Procedure: vNOTES Hysterectomy — Transluminal endoscopic hysterectomy is performed through a vaginal natural opening via transvaginal access using a self-adhering vaginal port.
  Arms: vNOTES Group
Procedure: Total Laparoscopic Hysterectomy — It is a conventional total laparoscopic hysterectomy performed using an umbilical cord port and two accessory trocars.
  Arms: TLH Group

SUMMARY:
This study is a prospective, randomized controlled trial comparing two different minimally invasive hysterectomy techniques: vaginal natural orifice transluminal endoscopic surgery (vNOTES) and conventional total laparoscopic hysterectomy (TLH). The aim is to evaluate whether vNOTES provides better postoperative comfort and recovery by reducing pain, lowering opioid analgesic requirements, and improving early recovery outcomes.

Approximately 80 women undergoing elective hysterectomy will be randomly assigned to either vNOTES or TLH. All surgeries will be performed under standardized general anesthesia by the same experienced surgical team. Postoperative pain management will follow an identical protocol for all patients.

Primary outcomes include postoperative pain scores (at 12 and 24 hours) and total opioid consumption. Secondary outcomes include Quality of Recovery-15 (QoR-15) scores, fatigue scores, time to first mobilization, time to first flatus, and length of hospital stay. The results of this study may help identify which hysterectomy technique offers better patient-centered recovery and postoperative comfort.

DETAILED DESCRIPTION:
This study is a single-center, prospective, randomized controlled clinical trial designed to compare two minimally invasive hysterectomy techniques: vaginal natural orifice transluminal endoscopic surgery (vNOTES) and conventional total laparoscopic hysterectomy (TLH). The aim is to determine whether vNOTES offers advantages in postoperative pain control, opioid requirements, and early recovery outcomes by eliminating abdominal wall incisions and reducing pneumoperitoneum-related physiological effects.

Eligible ASA I-II female patients aged 18-75 scheduled for elective hysterectomy are randomly assigned in a 1:1 ratio to the vNOTES or TLH group using a computer-generated sequence with sealed opaque envelopes for allocation concealment. All procedures are performed by the same experienced surgical and anesthesia team using a standardized general anesthesia protocol. Postoperative analgesia and recovery care are identical for both groups to ensure uniformity of perioperative management.

In the vNOTES group, hysterectomy is performed via transvaginal access using a self-retaining vaginal port, with pneumoperitoneum pressure kept at or below 15 mmHg. In the TLH group, a standard laparoscopic approach using a 10 mm umbilical port and two 5 mm accessory trocars is applied, with pneumoperitoneum maintained between 12-15 mmHg. Trendelenburg positioning is used in both techniques but is expected to be less steep and shorter in duration in the vNOTES group.

Outcome assessment is conducted by nurses and clinicians blinded to group allocation. Primary endpoints include postoperative pain scores at 12 and 24 hours (measured using a 0-10 Visual Analog Scale) and total opioid consumption within the first 24 hours. Secondary endpoints include Quality of Recovery-15 (QoR-15) scores, Fatigue Assessment Scale (FAS) scores, time to first mobilization, time to first flatus, length of hospital stay, and postoperative complications such as nausea/vomiting, shoulder pain, and respiratory discomfort. The study is powered based on a one-tailed hypothesis expecting lower postoperative discomfort in the vNOTES group.

The findings of this trial may help clarify whether vNOTES provides superior postoperative comfort and enhanced recovery compared to standard laparoscopic hysterectomy, contributing evidence to guide technique selection in minimally invasive gynecologic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18 to 75 years
* ASA physical status I-II
* Scheduled for elective laparoscopic hysterectomy (benign indications such as myoma uteri, adenomyosis, endometrial hyperplasia)
* Able to understand study procedures and provide written informed consent
* Able to complete postoperative questionnaires (QoR-15 and Fatigue Assessment Scale)

Exclusion Criteria:

* ASA III-IV status
* Severe cardiopulmonary disease or contraindication to general anesthesia
* Coagulopathy or bleeding disorders
* Active pelvic infection
* History of extensive pelvic or abdominal surgery complicating minimally invasive access
* Cognitive impairment or inability to complete questionnaires
* Conversion to laparotomy
* Known allergy or intolerance to study medications (paracetamol, tramadol)

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2026-01-08 (Actual); Primary Completion 2026-02-25 (Estimated); Study Completion 2026-02-26 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain Intensity (NRS) | At 12 and 24 hours postoperatively
  Postoperative pain intensity will be assessed using the 0-10 Numeric Rating Scale (NRS), where 0 indicates no pain and 10 indicates the worst imaginable pain.

SECONDARY OUTCOMES:
Need for Rescue Analgesia Within 24 Hours | First 24 postoperative hours
  The proportion of patients requiring rescue analgesia (intravenous tramadol 100 mg) after the standard regimen (paracetamol intravenously every 8 hours) will be recorded along with the number of rescue doses per patient.
Time to First Mobilization | From the end of surgery until the first ambulation out of bed, assessed up to 48 hours postoperatively.
  Time from the end of surgery to the first ambulation out of bed will be recorded in hours.
Time to First Flatus | Time Frame: From the end of surgery until the first passage of flatus, assessed during the postoperative hospital stay, up to 7 days postoperatively or until hospital discharge, whichever comes first.
  Time from the end of surgery to the first passage of flatus will be recorded in hours as an indicator of return of bowel function.
Length of Postoperative Hospital Stay | Time Frame: From the day of surgery until hospital discharge, assessed up to 30 days postoperatively or until discharge, whichever comes first.
  Length of stay will be calculated as the number of days from the day of surgery to the day of hospital discharge.
Change in QoR-15 Score from Baseline to 24 Hours | Time Frame: Preoperative (within 24 hours before surgery) and 24 hours postoperatively
  The Quality of Recovery-15 (QoR-15) questionnaire (total score 0-150; higher scores indicate better recovery) will be administered preoperatively and at 24 hours postoperatively. The primary analysis will focus on the change in total score from baseline to 24 hours.
Change in Fatigue Assessment Scale (FAS) Score from Baseline to 24 Hours | Preoperative (within 24 hours before surgery) and 24 hours postoperatively
  Fatigue will be evaluated using the Fatigue Assessment Scale (FAS; total score 10-50, higher scores indicate greater fatigue). The change in total score from baseline to 24 hours will be analyzed.
Postoperative Nausea and Vomiting (PONV) | During the first 24 hours postoperatively
  Postoperative nausea and vomiting will be recorded. Nausea severity will be assessed using a 0-10 Numeric Rating Scale (NRS), where 0 indicates no nausea and 10 indicates the worst imaginable nausea. Rescue antiemetic therapy will be administered if nausea severity is ≥4 or if vomiting occurs, and the need for rescue antiemetic treatment will be documented.
Estimated Intraoperative Blood Loss | During surgery
  Estimated blood loss (EBL) will be calculated based on the volume of blood collected in the suction canister after subtraction of irrigation fluids, combined with visual estimation of blood absorbed by surgical sponges, as recorded in the anesthesia chart.
Postoperative Hemoglobin Decrease | From preoperative baseline to 24 hours postoperatively
  Hemoglobin decrease will be calculated as the difference between preoperative hemoglobin level and postoperative hemoglobin level measured at 24 hours after surgery.
Perioperative Blood Transfusion Requirement | During surgery and up to 24 hours postoperatively
  The requirement for perioperative blood transfusion will be recorded as the administration of any packed red blood cells during surgery or within the first 24 hours postoperatively.
Postoperative Delirium and Acute Cognitive Dysfunction | Within the first 24 hours postoperatively
  Postoperative delirium and acute cognitive dysfunction will be assessed using the 4AT (4 'A's Test) screening tool within the first 24 hours after surgery. The 4AT evaluates four domains:
  1. Alertness (level of arousal),
  2. AMT4 (abbreviated mental test: age, date of birth, place, and current year),
  3. Attention (months of the year backwards),
  4. Acute change or fluctuating course.
  Scores range from 0 to 12, with 0 indicating normal cognition, 1-3 suggesting possible cognitive impairment, and ≥4 indicating probable delirium. The incidence of postoperative delirium (4AT ≥4) and acute cognitive dysfunction (4AT ≥1) will be recorded and compared between the vNOTES and TLH groups.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Acil, M.D., Principal Investigator — Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Locations (1):
- Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital, Diyarbakır, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fang S, Xia Y, Jin J, Zhang J, Lu L. Comparison of Surgical Outcomes Between Vaginally Assisted NOTES Hysterectomy and Laparoscopic Hysterectomy in Primary Hospitals: A Prospective Cohort Study. J Invest Surg. 2025 Dec;38(1):2515054. doi: 10.1080/08941939.2025.2515054. Epub 2025 Jun 10. PMID 40492370